CLINICAL TRIAL: NCT06811467
Title: Suicidal Ideation in Hereditary Angioedema
Brief Title: Suicide Ideation in Hereditary Angioedema
Acronym: HAE-SAFE
Status: Not yet recruiting | Type: Observational
Sponsor: Ivan Cherrez Ojeda (Other)
Responsible Party: Sponsor-Investigator, Ivan Cherrez Ojeda, Adjunct Professor, Charite University, Berlin, Germany
Organization: Charite University, Berlin, Germany (Other)
Other Study IDs: 2022-006
Record Dates: First submitted 2025-01-31; First posted 2025-02-06 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Hereditary Angioedema (HAE); Suicidal Ideation; Cardiovascular Risk
Keywords: Hereditary Angioedema; Suicidal ideation; TyG-BMI; cardiovascular risk
MeSH Terms: conditions — Angioedemas, Hereditary; Suicidal Ideation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- HAE-SAFE 1: Patients with a diagnosis of hereditary angioedema confirmed by decreased C1-INH levels and/or decreased C1-INH activity or genomic sequencing

SUMMARY:
This study focuses on patients with Hereditary Angioedema (HAE) to better understand how mental health affects overall well-being. Through a questionnaire, the investigators will assess the presence of suicidal thoughts, anxiety, and depression, as well as cardiovascular risk markers. By analyzing these factors together, the investigators aim to identify possible links between mental health and heart health in people with HAE. This research will help improve care strategies and highlight the importance of mental well-being in managing HAE.

DETAILED DESCRIPTION:
This observational study focuses on patients with Hereditary Angioedema (HAE) to explore the impact of mental health on overall well-being. Through a questionnaire, the investigators aim to assess not only the presence but also the severity of suicidal thoughts, as well as symptoms of anxiety and depression. Additionally, the investigators will evaluate how these mental health factors relate to disease variables such as HAE control, disease activity, and quality of life.

Beyond mental health, the investigators also seek to understand its connection to cardiovascular risk factors. By measuring triglycerides, glucose levels, and body mass index (BMI), the investigators aim to explore whether patients with higher suicide risk also face increased heart health risks. This research will help improve patient care by emphasizing the importance of both mental and physical health in managing HAE. After identifying patients with high risk of suicide ideation the investigators will conduct a folow-up study after patients have received mental health interventions and how evaluate how treatment can determine better HAE outcomes. With these resuts the investigators expect to attract the attention of the international scientific community to increase early detection and effective solutions to prevent suicide.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of hereditary angioedema
* Over the age of 18

Exclusion Criteria:

* Patients with intellectual disability
* Refusal to participate in the study
* Patients with acquired C1-INH deficiency
* Patients with other dermatological diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a confirmed diagnosis of hereditary angioedema who are treated at specialized centers in Latin America
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Presence of suicide ideation severity as assessed by the Suicidal Ideation Attributes Scale (SIDAS) | Day 1
  SIDAS measures five attributes of suicidal thoughts. Each attribute is scored on a 10-point scale, with total SIDAS scores ranging from 0 to 50. A score of 0= No ideation, 1-20= Low ideation, 21-50= High ideation .

SECONDARY OUTCOMES:
Number of participant with an increased triglyceride glucose-body mass (TyG-BMI) index | In the previous 12 weeks or up to 12 weeks after enrollment
  The TyG-BMI index will be obtained using the following formula: ln[TG (mg/dL) × FPG (mg/dL)/2] × BMI (kg/m^2), where TG represents for triglycerides and FBG represents for fasting blood glucose.
Number of patients with uncontrolled disease as assessed by the Angioedema Control Test (AECT) | Day 1
  A cut-off value of 10 points is used to differentiate patients with poor controlled angioedema from those with well-controlled disease
Number of patients with severe disease as assessed by the Hereditary Angioedema Activity Score: HAE-AS | Day 1
  A total score of 12 points will be used as a cutoff for severe disease
Number of patients with anxiety or depression as assessed by the Hospital Anxiety and Depression Scale (HADS) | Day 1
  HADS is a fourteen-item scale with seven items each for anxiety and depression subscales. Scoring for each item ranges from zero to three. A subscale score >8 denotes anxiety or depression.

IPD SHARING:
Plan to Share IPD: No
Data will be made available upon reasonable request to the principal investigato